CLINICAL TRIAL: NCT03876119
Title: CHemical OptImization of Cerebral Embolectomy in Patients With Acute Stroke Treated With Mechanical Thrombectomy (CHOICE) Trial
Brief Title: Intraarterial Alteplase Versus Placebo After Mechanical Thrombectomy
Acronym: CHOICE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Fundació La Marató de TV3 (Other); Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Principal Investigator, Angel Chamorro, M.D., Ph.D., Director, Comprehensive Stroke Center, Hospital Clinic Barcelona. Professor of Neurology, University of Barcelona., Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHOICE
Record Dates: First submitted 2019-03-12; First posted 2019-03-15 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Stroke, Acute
Keywords: Mechanical Thrombectomy; Recanalization; Reperfusion
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, placebo-controlled, double blind, phase 2b trial of acute stroke patients treated with MT, in which two therapies are compared: rt-PA or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The solutions of alteplase or placebo are limpid, transparent and colorless. Alteplase (Actilyse 10 mg powder and solvent for solution for injection and infusion) and placebo will be provided in kind by Boëhringer Ingelheim. The secondary conditioning of the investigation treatment will be performed by Alcura Health Spain S.A.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intraarterial alteplase (Experimental): All the patients will be given a 15 minutes IA infusion of alteplase (Actylise®) at a drug concentration of 1.0 mg/ml. At 15 minutes of IA treatment onset, the infusion will be stopped and the angiographic score assessed. If the angiographic score is improved compared with the baseline score the procedure is terminated, otherwise a new angiographic series will be repeated in 10 minutes before the end of the procedure in front and profile projections.
  Study drug will be prepared according to the following steps:
  1. Dilute 3 vials of 10 mgs (alteplase) in 30 cc of sterile water for injection (SWI), to attain a 30 cc solution at a concentration of 1mg/ml
  2. Calculate the volume of cc of infusion and therefore the total dose as per the formula: (Patient's weight in Kgs multiplied by 0.225)
  Interventions: Drug: Intraarterial alteplase
- Placebo (Placebo Comparator): The placebo will consist of a lyophilized white powder containing 0.2 mol/L arginine phosphate, 0.01% polysorbate 80, and pH 7.4 after reconstitution.
  Study drug will be prepared according to the following steps:
  1. Dilute 3 vials of 10 mgs (placebo) in 30 cc of sterile water for injection (SWI), to attain a 30 cc solution at a concentration of 1mg/ml
  2. Calculate the volume of cc of infusion and therefore the total dose as per the formula: (Patient's weight in Kgs multiplied by 0.225)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Intraarterial alteplase — See arm/group descriptions.
  Other Names: Intraarterial alteplase recombinant tissue plasminogen activator (rTPA)
  Arms: Intraarterial alteplase
Drug: Placebo — See arm/group descriptions.
  Arms: Placebo

SUMMARY:
Multicenter, randomized, placebo-controlled, double blind, phase 2b trial of acute stroke patients treated with mechanical thrombectomy (MT), in which two therapies are compared: rt-PA or placebo. Allocation at each center will account for 1 stratum: use of alteplase (yes vs. no) before MT. Subjects will be followed up to 90 days post-randomization.

DETAILED DESCRIPTION:
The study objective is to evaluate whether rt-PA is safe and efficient as an add-on to mechanical thrombectomy in patients with acute ischemic stroke and complete or near-complete recanalization of a proximal vessel occlusion and successful brain reperfusion on cerebral angiogram (corresponding to mTICI score 2b/3) The study is a multicenter, randomized, placebo-controlled, double blind, phase 2b trial of acute stroke patients treated with MT, in which two therapies are compared: rt-PA or placebo. Allocation at each center will account for 1 stratum: use of alteplase (yes vs. no) before MT. Subjects will be followed up to 90 days post-randomization

Patients will be enrolled in the angiosuit by interventionalists or neurologists once a mTICI 2b/3 is confirmed on cerebral angiography. The primary outcome is the proportion of patients with a mRS 0 to 1 at 90 days. A sample size of 100 patients per treatment arm in a 1:1 allocation will have at least 80% statistical power for the primary outcome (mRS with 0-1 score values) assuming a rate of 40% in the control arm and a 21% benefit in the experimental arm (odds ratio (OR) of 2.33) for a 5% two-sided type I error. This sample size will also guarantee the study power for that relative treatment benefit even if the success rate in the control group rises up to ≈56%. No study losses are accounted for since all randomised patients will be included in the analysis.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Patients with symptomatic large vessel occlusion (LVO) in the anterior, middle or posterior cerebral artery treated with MT resulting in an mTICI score 2b/3 at end of the procedure.. Patients with an mTICI score 2b/3 on the diagnostic cerebral angiography before the onset of MT are also eligible for the study.
2. Estimated delay to onset of rescue intraarterial rt-PA administration <24 hours from symptom onset, defined as the point in time the patient was last seen well
3. No significant pre-stroke functional disability (modified Rankin scale 0-1), or mRS >1 that according to the investigator is not related to neurological disease (i.e. amputation, blindness)
4. Age ≥18
5. ASPECTS >6 on non-contrast CT (NCCT) scan or MRI if symptoms lasting <4.5 hours or ASPECTS >6 on CT-Perfusion (CTP) or DWI-MRI if symptoms >4.5 <24 hours.
6. Informed consent obtained from patient or acceptable patient surrogate

EXCLUSION CRITERIA:

1. NIHSS score on admission >25
2. Contraindication to IV t-PA as per local national guidelines (except time to therapy)
3. Use of carotid artery stents during the endovascular procedure requiring dual antiplatelet therapy during the first 24h
4. Female who is pregnant or lactating or has a positive pregnancy test at time of admission
5. Current participation in another investigation drug or device treatment study (except observational study i.e.: RACECAT or clinical trials not testing new medical devices or new drugs i.e.IMAGECAT)
6. Known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency
7. Known coagulopathy, INR > 1.7 or use of novel anticoagulants < 48h from symptom onset
8. Platelets < 50,000
9. Renal Failure as defined by a serum creatinine > 3.0 mg/dl (or 265.2 μmol/l) or glomerular Filtration Rate [GFR] < 30
10. Subject who requires hemodialysis or peritoneal dialysis, or who have a contraindication to an angiogram for whatever reason
11. Any hemorrhage on CT/MRI
12. Clinical presentation suggests a subarachnoid hemorrhage, even if initial CT or MRI scan is normal
13. Suspicion of aortic dissection
14. Subject currently uses or has a recent history of illicit drug(s) or abuses alcohol
15. History of life threatening allergy (more than rash) to contrast medium
16. SBP >185 mmHg or DBP >110 mmHg refractory to treatment
17. Serious, advanced, terminal illness with anticipated life expectancy < 6 months
18. Pre-existing neurological or psychiatric disease that would confound evaluation
19. Presumed vasculitis or septic embolization
20. Unlikely to be available for 90-day follow-up (e.g. no fixed home address, visitor from overseas)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Good outcome at 90 days | Day 90 after treatment.
  The primary outcome will be the proportion of patients with a mRS 0 to 1 at 90 days

SECONDARY OUTCOMES:
Shift analysis of the 90-day modified Rankin Scale (mRS). | Day 90 after treatment.
  The shift analysis of the modified Rankin Scale (mRS), at day 90. The mRS at 90 days will be analyzed using a proportional odds model (POM) that combine into single worst rank the last two categories (5: severe incapacity and 6: death).
Infarct expansion ratio. | 48 (+/- 24h) hours of stroke
  Infarct Expansion Ratio on DWI-MRI (continuous variable), at 48h (+/- 24h) of stroke
Rate of infarct expansion at 24 hours. | 48 (+/- 24h) hours of stroke
  Proportion of patients with/without infarct expansion (dichotomous variable).
Final infarct volume. | 48 (+/- 24h) hours of stroke
  Infarction Volume on Diffusion Weighted Imaging (Magnetic Resonance Imaging) at 48h (+/- 24h) of stroke onset
Angiographic improvement on the Arterial Occlusive Lesion (AOL) scale | 10 minutes after treatment
  Proportion of patients with angiographic improvement on the Arterial Occlusive Lesion (AOL) scale. AOL describes arterial patency at the site of occlusion based on the degree of luminal opening (none, partial, or complete) with further qualification based simply on the presence (grades 2 or 3) or absence (grades 0 or 1) of any downstream flow.
TERTIARY OUTCOME: Barthel Scale at day 90 | Day 90 after treatment.
  Barthel Scale score of 95 to 100, at day 90
TERTIARY OUTCOME: Ischemic worsening within 72 hours os stroke onset | 72 hours of stroke onset
  Ischemic worsening (≥ 4 points in the NIHSS score) within 72 hours of stroke onset not attributable to stroke recurrence
TERTIARY OUTCOME: Quality of life measured at 90 days | Day 90 after treatment.
  Quality of life measured with the EuroQol Group 5-Dimension Self-Report Questionnaire (EQ-5D-3L) at 90 days

OTHER OUTCOMES:
Proportion of patients with improved mTICI 2b score | 10 minutes after treatment
  Proportion of patients with improved mTICI 2b score
  1. IV Alteplase use on admission (yes versus no)
  2. MT started within 7.3h of symptoms onset versus MT started between 7.4h and 24h.
  3. Admission serum glucose concentration≤100 mg/dL versus >100 mg/dL
  4. Males vs. Females
  5. Baseline angiographic score mTICI2b brain reperfusion versus baseline angiographic score eTICI2c/3 brain reperfusion.

CONTACTS AND LOCATIONS:
Overall Officials: Angel Chamorro, MD, PhD, Study Chair — Comprehensive Stroke Center, Hospital Clinic Barcelona.; Arturo Renú, MD, PhD, Principal Investigator — Comprehensive Stroke Center, Hospital Clinic Barcelona.; Marián Muchada, MD, PhD, Principal Investigator — Hospital Universitario de Vall d'Hebrón; Elisa Cuadrado, MD, PhD, Principal Investigator — Hospital del Mar; Anna Ramos, MD, Principal Investigator — Germans Trias i Pujol Hospital; Pol Camps, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Pere Cardona, MD, PhD, Principal Investigator — Hospital Universitari de Bellvitge; Mikel Terceño, MD, Principal Investigator — University Hospital of Girona Dr. Josep Trueta
Locations (7):
- Spain (7):
  - Germans Trias i Pujol Hospital, Badalona
  - Hospital Clinic of Barcelona, Barcelona
  - Hospital del Mar, Barcelona
  - Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Josep Trueta (HJT), Girona

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data on outcome measures will be published along with the main results of the trial.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available after publication of main study results.
Access Criteria: The IPD will be available from the Sponsor of the trial on reasonable request.

REFERENCES:
- [Background] Chamorro A, Blasco J, Lopez A, Amaro S, Roman LS, Llull L, Renu A, Rudilosso S, Laredo C, Obach V, Urra X, Planas AM, Leira EC, Macho J. Complete reperfusion is required for maximal benefits of mechanical thrombectomy in stroke patients. Sci Rep. 2017 Sep 14;7(1):11636. doi: 10.1038/s41598-017-11946-y. PMID 28912596
- [Background] Davalos A, Cobo E, Molina CA, Chamorro A, de Miquel MA, Roman LS, Serena J, Lopez-Cancio E, Ribo M, Millan M, Urra X, Cardona P, Tomasello A, Castano C, Blasco J, Aja L, Rubiera M, Gomis M, Renu A, Lara B, Marti-Fabregas J, Jankowitz B, Cerda N, Jovin TG; REVASCAT Trial Investigators. Safety and efficacy of thrombectomy in acute ischaemic stroke (REVASCAT): 1-year follow-up of a randomised open-label trial. Lancet Neurol. 2017 May;16(5):369-376. doi: 10.1016/S1474-4422(17)30047-9. Epub 2017 Mar 16. PMID 28318984
- [Background] Jovin TG, Chamorro A, Cobo E, de Miquel MA, Molina CA, Rovira A, San Roman L, Serena J, Abilleira S, Ribo M, Millan M, Urra X, Cardona P, Lopez-Cancio E, Tomasello A, Castano C, Blasco J, Aja L, Dorado L, Quesada H, Rubiera M, Hernandez-Perez M, Goyal M, Demchuk AM, von Kummer R, Gallofre M, Davalos A; REVASCAT Trial Investigators. Thrombectomy within 8 hours after symptom onset in ischemic stroke. N Engl J Med. 2015 Jun 11;372(24):2296-306. doi: 10.1056/NEJMoa1503780. Epub 2015 Apr 17. PMID 25882510
- [Background] Renu A, Blasco J, Millan M, Marti-Fabregas J, Cardona P, Oleaga L, Macho J, Molina C, Roquer J, Amaro S, Davalos A, Zarco F, Laredo C, Tomasello A, Guimaraens L, Barranco R, Castano C, Vivas E, Ramos A, Lopez-Rueda A, Urra X, Muchada M, Cuadrado-Godia E, Camps-Renom P, Roman LS, Rios J, Leira EC, Jovin T, Torres F, Chamorro A; CHOICE Investigators. The Chemical Optimization of Cerebral Embolectomy trial: Study protocol. Int J Stroke. 2021 Jan;16(1):110-116. doi: 10.1177/1747493019895656. Epub 2019 Dec 18. PMID 31852410
- [Result] Renu A, Millan M, San Roman L, Blasco J, Marti-Fabregas J, Terceno M, Amaro S, Serena J, Urra X, Laredo C, Barranco R, Camps-Renom P, Zarco F, Oleaga L, Cardona P, Castano C, Macho J, Cuadrado-Godia E, Vivas E, Lopez-Rueda A, Guimaraens L, Ramos-Pachon A, Roquer J, Muchada M, Tomasello A, Davalos A, Torres F, Chamorro A; CHOICE Investigators. Effect of Intra-arterial Alteplase vs Placebo Following Successful Thrombectomy on Functional Outcomes in Patients With Large Vessel Occlusion Acute Ischemic Stroke: The CHOICE Randomized Clinical Trial. JAMA. 2022 Mar 1;327(9):826-835. doi: 10.1001/jama.2022.1645. PMID 35143603

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-28): https://cdn.clinicaltrials.gov/large-docs/19/NCT03876119/Prot_SAP_001.pdf